CLINICAL TRIAL: NCT07056686
Title: Early Detection of Breast Cancer Among Women in the Middle Region of Syria
Brief Title: Early Detection of Breast Cancer Among Syrian Women
Status: Enrolling by invitation | Type: Observational
Sponsor: Al-Hawash Private University (Other)
Responsible Party: Sponsor
Other Study IDs: 01-05-2025
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Detection
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mammogram — Each patient will undergo a mammogram and echo of the breast used to detect early signs of cancer, such as tumors or calcifications, before symptoms appear.

SUMMARY:
The goal of this observational study is to evaluate breast cancer awareness, screening practices, and barriers to early detection among women in the middle region of Syria. The main questions it aims to answer are:

1. What is the level of awareness among women in this region regarding breast cancer symptoms and risk factors.
2. How do women practice breast self-examination and professional screenings.
3. What barriers prevent women from seeking early detection and treatment? Participants will complete a survey assessing their knowledge, behaviors, and challenges related to breast cancer screening. The findings will inform public health interventions to improve awareness and early detection practices.

ELIGIBILITY:
Women aged 18 years and older residing in the middle region of Syria.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in the middle reagon between 18-65 years old
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with early signs of breast cancer | From Participant enrolment to the end of the study at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hawash Private University, Homs, Syria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT07056686/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT07056686/ICF_001.pdf